CLINICAL TRIAL: NCT03924336
Title: Evaluation of CAL Gain Following Treatment of Intraosseous Defects With A-PRF+ Compared to Open Flap Debridement in Patients With Stage III Periodontitis: A Randomized Clinical Trial
Brief Title: The Effect of A-PRF+ Versus Open Flap Debridement in the Treatment of Patients With Stage III Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasser Ali Abdu, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01003884812
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-12

CONDITIONS: Intrabony Periodontal Defect
Keywords: stage 3 periodontitis; A-PRF; Advanced platelet rich fibrin; open flap debridement; OFD; 2-wall intraosseous defect; 3-wall intraosseous defect
MeSH Terms: conditions — Periodontitis | interventions — Single Person

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the type of intervention only the outcome assessor and the statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced- platelets rich fibrin plus with open flap debridement (Experimental): Mucoperiosteal flaps will be elevated using an intrasulcular incision buccally and palatally or lingually. Then the defects will be thoroughly debrided using curettes and ultrasonic scalers. The clinical measurements will be then recorded. After debridement and intraoperative recordings, A-PRF+ of the required size will be filled into the intraosseous defect, the mucoperiosteal flaps will be repositioned and secured in place using 4-0 silk sutures
  Interventions: Procedure: Advanced- platelets rich fibrin (A-PRF+) + Open flap debridement (OFD)
- Open flap debridement (OFD) (Active Comparator): Mucoperiosteal flaps will be elevated using an intrasulcular incision buccally and palatally or lingually. Then the defects will be thoroughly debrided using curettes and ultrasonic scalers. The clinical measurements will be then recorded. After debridement and intraoperative recordings, The interrupted sutures using 4-0 silk sutures will be placed to reposition the flaps.
  Interventions: Procedure: Open flap debridement (OFD) alone

INTERVENTIONS:
Procedure: Advanced- platelets rich fibrin (A-PRF+) + Open flap debridement (OFD) — Elevation of flap.Thorough debridement of the defects using curettes and ultrasonic scalers. Clinical measurements will be then recorded , A-PRF+ of the required size will be filled into the intraosseous defect. The mucoperiosteal flaps will be repositioned and secured in place using4-0 silk sutures
  Arms: Advanced- platelets rich fibrin plus with open flap debridement
Procedure: Open flap debridement (OFD) alone — Elevation of flap.Thorough debridement of the defects using curettes and ultrasonic scalers. Clinical measurements will be then recorded. After debridement and intraoperative recordings, interrupted sutures using 4-0 silk sutures will be placed to reposition the flaps.
  Arms: Open flap debridement (OFD)

SUMMARY:
To assess the effectiveness of advanced PRF+ as compared to open flap debridement in treatment of periodontal intraosseous defects in stage III periodontitis patients.

DETAILED DESCRIPTION:
The application of platelet concentrates characterized by high concentrations of platelets and growth factors have been applied and investigated as possible periodontal regenerative therapy. The application of platelet rich fibrin in management of intraosseous and furcation defects produce more favorable outcome compared to open flap debridement.

A-PRF+ represents the latest generation of platelet concentrates that could provide sustained and increased release of growth factors and could serve as an autologous cost-effective membrane in periodontal tissue regeneration procedures

ELIGIBILITY:
Inclusion Criteria:

* Stage III periodontitis patient having at least one tooth with 2-wall, 3-wall, or combined 2- to 3-wall intraosseous defect ≥ 3 mm in depth (assessed by bone sounding, radiographic examination) with clinical attachment level (CAL) ≥ 5mm and pocket depth (PD) ≥ 6 mm.
* Defect not extending to a root furcation area
* Non-smokers.
* No history of intake of medications affecting the periodontium in the previous 6 months.
* Able to sign an informed consent form.
* Patients age between 18 and 60 years old.
* Patients who are cooperative, motivated, and hygiene conscious.
* Systemically free according to Cornell Medical Index (Broadbent, 1951).

Exclusion Criteria:

* Pregnancy or breast feeding
* The presence of an orthodontic appliance
* Teeth mobility greater than grade I

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

PRIMARY OUTCOMES:
Clinical Attachment Level (CAL) gain | Change from Baseline Clinical Attachment Level (CAL) at 9 months
  Clinical Attachment Level (CAL) will be measured from the cemento enamel junction (CEJ) to the bottom of the gingival sulcus/periodontal pocket using University of North Carolina (UNC) periodontal probe at six sites per tooth

SECONDARY OUTCOMES:
Probing Depth (PD) | Probing Depth will be measured at base line,3,6, and 9 months postoperative
  Probing Depth (PD) will be measured from the gingival margin to the bottom of the gingival sulcus/ periodontal pocket using University of North Carolina (UNC) periodontal probe at six sites per tooth
Radiographic defect fill | Radiographic defect fill will be measured at 6,9,months
  The depth of intrabony defect (IBD) will be measured from the alveolar bone crest to the base of the defect at baseline and after six months to detect the amount of bone fill Individually customized bite blocks and parallel-angle technique will be used to obtain standardized radiographs. Radiographs will be scanned and the radiographic (intrabony defect) IBD depth was measured by a computer-aided software program
Gingival Recession Depth (RD) | Gingival Recession Depth will be measured at base line,3,6, and 9 months postoperative
  Gingival Recession Depth (RD) will be measured from the cemento enamel junction (CEJ) to the most apical extension of the gingival margin using University of North Carolina (UNC) periodontal probe at six sites per tooth

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, Professor, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

REFERENCES:
- [Result] Cortellini P, Tonetti MS. Clinical concepts for regenerative therapy in intrabony defects. Periodontol 2000. 2015 Jun;68(1):282-307. doi: 10.1111/prd.12048. PMID 25867990
- [Result] Kobayashi E, Fluckiger L, Fujioka-Kobayashi M, Sawada K, Sculean A, Schaller B, Miron RJ. Comparative release of growth factors from PRP, PRF, and advanced-PRF. Clin Oral Investig. 2016 Dec;20(9):2353-2360. doi: 10.1007/s00784-016-1719-1. Epub 2016 Jan 25. PMID 26809431